CLINICAL TRIAL: NCT04840953
Title: Negative Pressure Therapy, Minimally Invasive and Accessible Technique in the Treatment of Massive Subcutaneous Emphysema in COVID-19 or Non Infected Critical Patients
Status: Completed | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Luis Sánchez Guillen, Colorrectal Surgeon, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: ENFIVAC
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Subcutaneous Emphysema; Covid19
MeSH Terms: conditions — Subcutaneous Emphysema; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vçac — VAC THERAPY vs SURGICAL DREINAGE

SUMMARY:
Background Numerous surgicals treatments have been described for the massive subcutaneous emphysema; however, some of these techniques cannot be carried out in a critical care unit and they are related with high morbidity and exposure in positive SARS COV-2 patients. More effective, less invasive and isolated procedures should be implemented.

Technique Negative pressure therapy (NPT) that can allow effective solving of massive subcutaneous emphysema in a short period (5 days) with a minimally invasive approach at the bedside in Covid-19 or non infected critical patients.

Conclusion NPT is an effective and low invasive strategy for the management of EES in critical patients with high risk of mortality.

ELIGIBILITY:
Inclusion Criteria:

* Subcutaneous emphysema that compromises ventilation

Exclusion Criteria:

* Declined Therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subcutaneous emphysema that compromises ventilation with or not SARS COV2 infection
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Resolution time of emphysema with negative pressure therapy | Days
  Days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No